CLINICAL TRIAL: NCT07407998
Title: Evaluation of Artificial Intelligence Models in Assigning American Society of Anesthesiologists Physical Status Classification in Preoperative Patients: A Prospective Observational Study
Brief Title: AI-Based ASA Classification in Preoperative Patients
Acronym: AI-Based ASA C
Status: Completed | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, eralp çevikkalp, assos proc., Bursa City Hospital
Other Study IDs: Bursa City Hospital 004
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Preoperative Risk Assessment; ASA Physical Status Classification
Keywords: Artificial Intelligence; Large Language Models; Preoperative Evaluation; ASA Classification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to evaluate the performance of multiple artificial intelligence-based large language models in assigning American Society of Anesthesiologists Physical Status (ASA-PS) classifications in adult preoperative patients. AI-generated ASA scores obtained using both prompted and unprompted clinical scenario inputs will be compared with assessments performed by experienced anesthesiologists. The agreement, accuracy, readability, and overall quality of AI outputs will be analyzed to determine the potential role of artificial intelligence in supporting preoperative risk stratification.

DETAILED DESCRIPTION:
The American Society of Anesthesiologists Physical Status (ASA-PS) classification is widely used for perioperative risk stratification but is subject to interobserver variability. Recent advances in artificial intelligence and large language models have introduced new opportunities for clinical decision support.

This prospective observational study includes adult patients undergoing routine preoperative anesthesia evaluation at Bursa City Hospital. Demographic data, medical history, comorbidities, functional capacity, laboratory findings, electrocardiography, chest imaging results, and planned surgical procedures are recorded to construct standardized clinical scenarios.

Multiple artificial intelligence models, including large language model-based systems, are provided with patient scenarios using both structured prompts and unstructured inputs. Each model assigns an ASA-PS classification and provides explanatory text. AI-generated classifications are compared with assessments performed independently by experienced anesthesiologists.

Primary outcomes include agreement and accuracy between AI-generated and clinician-assigned ASA classifications using Cohen's Kappa statistics. Secondary outcomes include readability assessment using the Ateşman Turkish Readability Index and response quality evaluation using the Global Quality Scale.

The study aims to explore whether artificial intelligence can improve standardization, objectivity, and efficiency in preoperative risk assessment while highlighting the strengths and limitations of current AI technologies in clinical anesthesia practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Undergoing routine preoperative anesthesia evaluation
* Classified as ASA Physical Status I-IV
* Availability of complete clinical data required for AI assessment

Exclusion Criteria:

* Patients younger than 18 years
* Refusal to participate
* Incomplete or missing clinical information

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients presenting for routine preoperative anesthesia assessment at Bursa City Hospital, including individuals with varying comorbidities and surgical risk profiles.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Agreement Between AI-Generated and Clinician-Assigned ASA Physical Status Classification | Preprocedural/Perioperative
  Level of agreement between artificial intelligence models and anesthesiologists in assigning ASA Physical Status classification measured using Cohen's Kappa coefficient

SECONDARY OUTCOMES:
Accuracy of AI Models in ASA Classification | Preprocedural/Perioperative
  Proportion of correct ASA Physical Status classifications generated by artificial intelligence models compared with anesthesiologist assessments
Readability of AI-Generated Clinical Responses | Preprocedural/Perioperative
  Readability scores of artificial intelligence-generated clinical responses assessed using the Ateşman Turkish Readability Index (range: 0-100), where higher scores indicate better readability.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient confidentiality and institutional data protection policies.